CLINICAL TRIAL: NCT06516965
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Efficacy and Safety Study of Povorcitinib in Participants With Prurigo Nodularis
Brief Title: A Study to Evaluate the Efficacy and Safety Study of Povorcitinib in Participants With Prurigo Nodularis (STOP-PN2)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCB54707-306; 2024-511881-35-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Prurigo Nodularis
Keywords: Prurigo nodularis; PN; INCB054707; chronic pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Povorcitinib Dose 1 (Experimental): Povorcitinib at the protocol-defined dose.
  Interventions: Drug: Povorcitinib
- Povorcitinib Dose 2 (Experimental): Povorcitinib at the protocol-defined dose.
  Interventions: Drug: Povorcitinib
- Placebo (Placebo Comparator): Placebo at the protocol-defined dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Povorcitinib — Oral Tablet
  Other Names: INCB054707
  Arms: Povorcitinib Dose 1; Povorcitinib Dose 2
Drug: Placebo — Oral Tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate effect of povorcitinib on itch and skin lesions in participants with prurigo nodularis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants 18 to 75 years of age.
* Clinical diagnosis of PN for at least 3 months prior to Screening visit.
* Pruritus, defined as an average Itch NRS score ≥ 7 during the 7 days prior to Day 1/Baseline.
* Total of ≥ 20 pruriginous lesions on ≥ 2 different body regions (both legs, and/or both arms, and/or trunk) at Screening and Day 1/Baseline.
* Documented history of treatment failure, demonstrated intolerance, or contraindication to a previous PN treatment.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Chronic pruritus due to a condition other than PN or neuropathic and psychogenic pruritus.
* Diagnosis of PN secondary to medications.
* Active AD lesions (signs and symptoms other than dry skin) within 3 months prior to Screening visit.
* Women who are pregnant (or are considering pregnancy) or breastfeeding.
* Medical history including thrombocytopenia, coagulopathy or platelet dysfunction; venous and arterial thrombosis, deep vein thrombosis, pulmonary embolism, stroke, moderate to severe heart failure, cerebrovascular accident, myocardial infarction, or other significant cardiovascular diseases; Q-wave interval abnormalities; disseminated herpes zoster or dermatomal herpes zoster; disseminated herpes simplex; chronic/recurrent infections; malignancies.
* Evidence of infection with TB, HBV, HCV or HIV.
* History of failure to any topical or systemic JAK or TYK2 inhibitor as treatment of PN or any inflammatory disease.
* Laboratory values outside of the protocol-defined ranges.

Other protocol-defined Inclusion/Exclusion Criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-10-19 (Estimated); Study Completion 2027-05-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving Itch NRS4 and IGA-CPG-S-TS at Week 24 | Week 24
  Defined as proportion of participants achieving a ≥ 4-point improvement [reduction] in Itch NRS score from baseline (Itch NRS4) and an IGA CPG-S score of 0 or 1 with a ≥ 2-grade improvement from baseline (IGA-CPG-S-TS).

SECONDARY OUTCOMES:
Proportion of participants achieving Itch NRS4 at Week 24 | Week 24
  Defined as percentage of participants that achieve a ≥ 4-point improvement (reduction) in Itch NRS score from baseline.
Proportion of participants achieving IGA-CPG-S-TS at Week 24 | Week 24
  Defined as percentage of participants that achieve IGA-CPG-S score of 0 or 1 with a ≥ 2 grade improvement from baseline.
Proportion of participants achieving Itch NRS4 at Week 4 | Week 4
  Defined as percentage of participants that achieve a ≥ 4-point improvement (reduction) in Itch NRS score from baseline.
Time to Itch NRS4 | Up to 52 Weeks
  Defined as time taken for the participant to achieve a ≥4 improvement in Itch NRS score from baseline.
Change from baseline in Itch NRS score at each postbaseline visit | Up to 52 weeks
  Itch will be measured using an NRS used to indicate the intensity of the worst itching over the past 24 hours using a 0 to 10 numeric rating scale, where "0" represents "no itching" and "10" represents "worst itching imaginable".
Percent change from baseline in NRS score at each postbaseline visit | Up to 52 weeks
  Itch will be measured using an NRS used to indicate the intensity of the worst itching over the past 24 hours using a 0 to 10 numeric rating scale, where "0" represents "no itching" and "10" represents "worst itching imaginable".
Proportion of participants achieving Itch NRS4 at each postbaseline visit | Up to 52 weeks
  Defined as percentage of participants that achieve a ≥ 4-point improvement in Itch NRS score from baseline.
Proportion of participants achieving IGA-CPG-S-TS at each postbaseline visit | Up to 52 weeks
  Defined as percentage of participants that achieve an IGA-CPG-S score of 0 or 1 with a ≥ 2 grade improvement from baseline.
Proportion of participants achieving Investigator's Global Assessment - Chronic Prurigo Activity (IGA-CPG-A) at each postbaseline visit | Up to 52 weeks
  Defined as percentage of participants that achieve an IGA-CPG-A score of 0 or 1 with a ≥ 2 grade improvement (reduction) from baseline.
Proportion of participants achieving ≥ 75% healed lesions in Prurigo Activity Score (PAS) at each postbaseline visit | Up to 52 weeks
  The modified PAS will be used in this study as defined by the protocol.
Proportion of participants achieving Itch NRS4 and IGA-CPG-S-TS at each postbaseline visit | Up to 52 weeks
  Defined as percentage of participants that achieve a ≥ 4-point improvement (reduction) in Itch NRS score and IGA-CPG-S score of 0 or 1 with a ≥ 2-grade improvement from baseline.
Change from baseline in Dermatology Life Quality Index (DLQI) score at each postbaseline visit. | Up to 52 weeks
  The DLQI is a simple, 10-question validated questionnaire to measure how much the skin problem has affected the participant over the previous 7 days.
Percent change from baseline in Dermatology Life Quality Index (DLQI) score at each postbaseline visit. | Up to 52 weeks
  The DLQI is a simple, 10-question validated questionnaire to measure how much the skin problem has affected the participant over the previous 7 days.
Proportion of participants with at least a 4-point decrease in DLQI score from baseline at each postbaseline visit for participants with DLQI score ≥ 4 at baseline | Up to 52 weeks
  Defined as percentage of participants with at least a 4-point decrease in DLQI score from baseline at each postbaseline visit for participants with DLQI score ≥ 4 at baseline.
Change from baseline in Skin Pain NRS score at each postbaseline visit | Up to 52 weeks
  Skin Pain NRS is an 11-point scale (0 to10) where 0 is "no pain" and 10 is the "worst pain imaginable".
Percent change from baseline in Skin Pain NRS score at each postbaseline visit | Up to 52 weeks
  Skin Pain NRS is an 11-point scale (0 to10) where 0 is "no pain" and 10 is the "worst pain imaginable".
Change from baseline in the Hospital Anxiety and Depression Scale (HADS) score at each postbasline visit | Up to 52 weeks
  HADS is a 14-item questionnaire that assesses the levels of anxiety and depression that a participant is currently experiencing. There are 7 questions each for measuring anxiety and for measuring depression, with 4 possible responses to each question (responses are scored as 0, 1, 2, or 3).
Percent change from baseline in the HADS score at each postbaseline visit | Up to 52 weeks
  HADS is a 14-item questionnaire that assesses the levels of anxiety and depression that a participant is currently experiencing. There are 7 questions each for measuring anxiety and for measuring depression, with 4 possible responses to each question (responses are scored as 0, 1, 2, or 3).
Change from baseline in EQ-5D-5L score at each postbaseline visit | Up to 52 weeks
  The EQ-5D-5L questionnaire is a standardized, validated instrument for use as a measure of health outcome.
Percent change from baseline in EQ-5D-5L score at each postbaseline visit | Up to 52 weeks
  The EQ-5D-5L questionnaire is a standardized, validated instrument for use as a measure of health outcome.
Change in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) score at each postbaseline visit | Up to 52 weeks
  The FACIT-F is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function over the past 7 days.
Percent change in FACIT-F score at each postbaseline visit | Up to 52 weeks
  The FACIT-F is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function over the past 7 days.
Proportion of participants with at least a ≥ 4-point increase in FACIT-F score at each postbaseline visit for participants with FACIT-F score ≤ 48 at baseline | Up to 52 weeks
  The FACIT-F is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function over the past 7 days.
Number of Participants with Treatment Emergent Adverse Events (TEAE) | Up to 52 weeks
  Defined as any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (120):
- United States (28):
  - Medical Dermatology Specialists Phoenix, Phoenix, Arizona
  - Investigate Md, Scottsdale, Arizona
  - First Oc Dermatology Research Inc, Fountain Valley, California
  - Clinical Science Institute Clinical Research Specialists Inc, Santa Monica, California
  - Center For Clinical and Cosmetic Research, Aventura, Florida
  - Clearlyderm Dermatology, Boca Raton, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Skin Care Research, Llc, Hollywood, Florida
  - Ziaderm Research, Llc, Miami, Florida
  - Nodal Medical Center, Llc, Tampa, Florida
  - Trueblue Clinical Research Moore Clinical Research, Inc McR Tampa Clinic Location, Tampa, Florida
  - Dermatology Specialists Research, Louisville, Kentucky
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Dermatology Associates Pc, Rockville, Maryland
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - Fivenson Dermatology, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Michigan Dermatology Institute, Waterford, Michigan
  - Allcutis Research, Llc, Portsmouth, New Hampshire
  - Schweiger Dermatology, Hackensack, New Jersey
  - OPTISKIN, New York, New York
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - Central Sooner Research, Oklahoma City, Oklahoma
  - Paddington Testing Co Inc, Philadelphia, Pennsylvania
  - Yardley Dermatology Associates, Yardley, Pennsylvania
  - Modern Research Associates Pllc, Dallas, Texas
  - University of Utah Midvalley Dermatology, Murray, Utah
  - Aesthetic General Dermatology of Seattle, Burien, Washington
- Australia (7):
  - Novatrials, Charlestown, New South Wales
  - Premier Specialists Pty Ltd, Kogarah, New South Wales
  - Skin & Cancer Foundation Australia, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland
  - The Alfred Hospital, Melbourne, Victoria
  - Fremantle Dermatology, Fremantle
- Belgium (5):
  - Az Sint-Jan Brugge Av, Bruges
  - Universitair Ziekenhuis Gent (Uz Gent), Ghent
  - Grand Hopital de Charleroi - Site Imtr, Gilly
  - Centre Hospitalier Universitaire (Chu) de Liege - Domaine Universitaire Du Sart Tilman, Liège
  - Universite Catholique de Louvain (Ucl) - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
- Canada (8):
  - Skin Physicians, Edmonton, Alberta
  - Alpha Research-Lucere Dermatology and Laser Clinic, Edmonton, Alberta
  - Simcoderm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Dermeffects, London, Ontario
  - North York Research Inc., Toronto, Ontario
  - Toronto Research Centre, Toronto, Ontario
  - Centre de Recherche Saint-Louis, Québec, Quebec
  - Skinsense Medical Research, Saskatoon, Saskatchewan
- Chile (3):
  - Centro Medico Skinmed Limitada, Santiago
  - Centro Internacional de Estudios Clinicos, Santiago
  - Clinical Research Chile Spa., Valdivia
- Czechia (3):
  - Clintrial S.R.O., Prague
  - Sanatorium Profesora Arenbergera, Prague
  - Sanixtra Prague, Prague
- Germany (14):
  - University Hospital Rwth Aachen, Aachen
  - Elbe Kliniken Buxtehude, Buxtehude
  - Drk Krankenhaus Chemnitz-Rabenstein, Chemnitz
  - Klinikum Darmstadt, Darmstadt
  - Rosenpark Research Gmbh, Darmstadt
  - University Hospital Carl Gustav Carus, Dresden
  - Klinikum Der Johann Wolfgang Goethe-Universitaet, Frankfurt am Main
  - Universitaetsmedizin Goettingen, Göttingen
  - Magdeburger Company For Medical Studies and Services Gmbh, Magdeburg
  - Dermatologische Gemeinschaftspraxis Dres. Quist, Mainz
  - Technischen Universitaet Muenchen, München
  - University Hospital Muenster, Münster
  - Klinikum Oldenburg Aor, Oldenburg
  - Hautarztpraxis Dr. Hoffmann, Witten
- Japan (19):
  - Tokyo Medical and Dental University Hospital, Faculty of Medicine, Bunkyō City
  - Tokyo Medical University Ibaraki Medical Center - Kasumigaura Campus (Tokyo Medical University Kasum, Inashiki-gun
  - Noguchi Dermatology Clinic, Kamimashiki-gun
  - Nippon Medical School Musashikosugi Hospital, Kawasaki-shi
  - University of Occupational and Environmental Health, Japan, Kitakyushu
  - Shimizu Dermatology Clinic, Kobe
  - Aoi Skin Clinic, Kumamoto
  - Dokkyo Medical University Saitama Medical Center, Minamikoshigaya
  - Central Japan International Medical Center, Minokamo
  - Niigata University Medical & Dental Hospital, Niigata
  - Medical Corporation Jun Dermatology Clinic, Osaka
  - Tanpopo Dermatology Clinic, Ōta-ku
  - Kume Derma Clinic, Sakai
  - Sapporo Skin Clinic, Sapporo
  - Tohoku University Hospital, Sendai
  - Tokyo Medical University Hospital, Shinjuku-ku
  - National Defence Medical College Hospital, Tokorozawa-shi
  - Queen'S Square Medical Facilities, Yokohama
  - Nomura Dermatology Clinic, Yokohama
- Poland (13):
  - Akk Medical Sp. Z O.O. - Centrum Medyczne Tu Sie Leczy, Gdansk
  - Care Clinic Sp. Z O.O., Katowice
  - Santa Familia Ptg Lodz, Lodz
  - Dermoklinika Centrum Medyczne S.C., M. Kierstan, J. Narbutt, A. Lesiak, Lodz
  - Luxderm Specjalistyczny Gabinet Dermatologiczny Prof. Dr. Hab. N. Med. Dorota Krasowska, Lublin
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski
  - Clinical Research Center Spolka Z Ograniczona Odpowiedzialnoscia Medic-R Spolka Komandytowa, Poznan
  - Uniwersytecki Szpital Kliniczny Im. Fryderyka Chopina W Rzeszowie, Rzeszów
  - Mics Centrum Medyczne Toruń, Torun
  - High-Med. Przychodnia Specjalistyczna, Warsaw
  - Panstwowy Instytut Medyczny Mswia, Warsaw
  - Royalderm Agnieszka Nawrocka, Warsaw
  - Cityclinic Przychodnia Lekarsko-Psychologiczna Matusiak Spolka Partnerska, Wroclaw
- Spain (13):
  - Hospital General Universitario Dr Balmis, Alicante
  - Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Clinico Universitario San Cecilio, Granada
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda
  - Hospital de Manis, Manises
  - Area Sanitaria de Santiago de Compostela Y Barbanza - Complejo Hospitalario Universitario de Santiag, Santiago de Compostela
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitari I Politecnic La Fe de Valencia - Instituto de Investigacion Sanitaria La Fe, Valencia
- United Kingdom (7):
  - The Dudley Group Nhs Foundation Trust, Dudley
  - Ipswich Hospital, East Suffolk and North Essex Nhs Foundation Trust, Ipswich
  - Broadgreen Hospital - Liverpool University Hospitals Nhs Foundation Trust, Liverpool
  - The Royal London Hospital - Barts Health Nhs Trust, London
  - Guy'S Hospital - Guy'S & St Thomas' Nhs Foundation Trust, London
  - Poole Hospital - University Hospitals Dorset Nhs Foundation Trust, Poole
  - Surrey and Sussex Healthcare Nhs Trust - East Surrey Hospital, Redhill

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A Study to Evaluate the Efficacy and Safety Study of Povorcitinib in Participants With Prurigo Nodularis (STOP-PN2) — https://incyteclinicaltrials.com/studies/incb54707-306